CLINICAL TRIAL: NCT00522691
Title: Efficacy of Sacral Nerve Stimulation Before Definitive Implantation: a Multicenter Randomized, Double Blind, Crossover Trial
Brief Title: Efficacy of Sacral Nerve Stimulation Before Definitive Implantation
Acronym: SNStest
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, PI, University of Lausanne Hospitals
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CHV120/07
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence; sacral nerve stimulation
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: sacral first (Experimental): Phase 1: sacral nerve stimulation crossover Phase 2 : sham stimulation
  Interventions: Procedure: sacral nerve stimulation
- B: sham first (Experimental): Phase 1: sham stimulation crossover Phase 2: sacral nerve stimulation
  Interventions: Procedure: sacral nerve stimulation

INTERVENTIONS:
Procedure: sacral nerve stimulation — sacral nerve stimulation for fecal incontinence

SUMMARY:
Sacral nerve stimulation (SNS) is an emerging treatment for patients with severe fecal incontinence. The test stimulation is minimally invasive, associated to low morbidity and relatively cheap. On the contrary, implantation of the definite stimulator is related to higher morbidity and considerable costs. A careful patent selection for definite implantation is therefore crucial. However, indication for implantation is actually based only on the subjective criteria reported in the patients´ diary only. Patients and care providers are likely to overestimate the real effect of SNS leading to an unjustified overuse of this expensive device. It is therefore necessary to evaluate real efficacy of SNS during the testing phase in a unbiased setting in order to avoid unnecessary morbidity and costs.

DETAILED DESCRIPTION:
Sacral nerve stimulation (SNS) is an emerging treatment for patients with severe faecal incontinence when conservative measures fail and surgical repair is not indicated. In a minimally-invasive approach and under local anaesthesia, an electrode is placed around sacral nerve root S2-4 and electrical stimulation is applied to the sacral spinal nerves. Effectiveness of SNS is definitively not only explained by placebo effect but the pathophysiologic mechanisms remain unclear. Suggested pathways include modulation of afferent nerve fibres and direct stimulation of the pelvic floor and anal sphincter muscle. After placement of the electrode, the patient is stimulated by an external stimulator for 1-3 weeks. During this period, the patient documents the number of faecal incontinence episodes or urgencies in a symptom diary. By convention, indication for permanent stimulation is based on a 50% reduction in the number of episodes. After a successful testing period, the permanent stimulator is implanted, generally in the upper gluteal region.

Previous studies report success rates up to 80%. The only randomized trial with a proper sample size evaluated the efficacy of SNS after definite implantation. In this study, 63% of the patients felt improved during the placebo period and might not really benefit from the device. The real success rate of SNS is therefore likely to be considerably lower. Efficacy of SNS during the testing phase has never been assessed in a blinded randomized study.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to SNS test for treatment of faecal incontinence after unsuccessful conservative (or surgical) treatment.

Exclusion criteria:

* Absence of informed consent.
* Patients not speaking french or german.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Primary success rate of SNS after 7 days. By convention this is assessed by >50% reduction in the number of episodes in the symptom diary. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hubner, MD, Principal Investigator — Visceral Surgery, University Lausanne, Switzerland; Jean-Claude Givel, Professor, Study Director — Visceral Surgery, University Lausanne, Switzerland; Nicolas Demartines, Professor, Study Chair — Visceral Surgery, University Lausanne, Switzerland
Locations (1):
- Visceral surgery, university hospital, Lausanne, Canton of Vaud, Switzerland